CLINICAL TRIAL: NCT05439408
Title: An Open Label, Balanced, Randomized, Two-Treatment, Two-Sequence, Four-Period, Full Replicate, Crossover, Single Dose, Oral Comparative Bioavailability Study of XS004 (Dasatinib) 100 mg Film-Coated Tablets, Formulation G of Xspray Pharma AB, Sweden, and SPRYCEL® (Dasatinib) 140 mg Film-Coated Tablets of Bristol-Myers Squibb Company, Princeton, NJ 08543 USA in Healthy, Adult Subjects Under Fasting Conditions
Brief Title: Comparative Bioavailability of XS004 (Dasatinib) Formulation G and SPRYCEL® (Dasatinib) in Healthy, Adult Subjects Under Fasting Conditions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Xspray Pharma AB (Industry)
Collaborators: QPS Bioserve India Pvt Limited (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: XS004-15
Record Dates: First submitted 2022-06-21; First posted 2022-06-30 (Actual); Last update posted 2022-06-30 (Actual); Status verified 2022-06

CONDITIONS: Biological Availability
MeSH Terms: interventions — Dasatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (8):
- XS004 - Period 1 (Experimental): At the clinic, after an overnight fast of at least 10 hours, a single oral dose of 100 mg tablet was administered to each participant in a sitting posture with about 240 mL of drinking water in the presence of the principal investigator and quality assurance personnel and in accordance with the randomization schedule.
  Interventions: Drug: Dasatinib ASD 100 mg
- SPRYCEL - Period 1 (Active Comparator): At the clinic, after an overnight fast of at least 10 hours, a single oral dose of 140 mg tablet was administered to each participant in a sitting posture with about 240 mL of drinking water in the presence of the principal investigator and quality assurance personnel, and in accordance with the randomization schedule.
  Interventions: Drug: Dasatinib 140 MG [Sprycel]
- XS004 - Period 2 (Experimental): At the clinic, after an overnight fast of at least 10 hours, a single oral dose of 100 mg tablet was administered to each participant in a sitting posture with about 240 mL of drinking water in the presence of the principal investigator and quality assurance personnel and in accordance with the randomization schedule.
  Interventions: Drug: Dasatinib ASD 100 mg
- SPRYCEL - Period 2 (Active Comparator): At the clinic, after an overnight fast of at least 10 hours, a single oral dose of 140 mg tablet was administered to each participant in a sitting posture with about 240 mL of drinking water in the presence of the principal investigator and quality assurance personnel, and in accordance with the randomization schedule.
  Interventions: Drug: Dasatinib 140 MG [Sprycel]
- XS004 - Period 3 (Experimental): At the clinic, after an overnight fast of at least 10 hours, a single oral dose of 100 mg tablet was administered to each participant in a sitting posture with about 240 mL of drinking water in the presence of the principal investigator and quality assurance personnel and in accordance with the randomization schedule.
  Interventions: Drug: Dasatinib ASD 100 mg
- SPRYCEL - Period 3 (Active Comparator): At the clinic, after an overnight fast of at least 10 hours, a single oral dose of 140 mg tablet was administered to each participant in a sitting posture with about 240 mL of drinking water in the presence of the principal investigator and quality assurance personnel, and in accordance with the randomization schedule.
  Interventions: Drug: Dasatinib 140 MG [Sprycel]
- XS004 - Period 4 (Experimental): At the clinic, after an overnight fast of at least 10 hours, a single oral dose of 100 mg tablet was administered to each participant in a sitting posture with about 240 mL of drinking water in the presence of the principal investigator and quality assurance personnel and in accordance with the randomization schedule.
  Interventions: Drug: Dasatinib ASD 100 mg
- SPRYCEL - Period 4 (Active Comparator): At the clinic, after an overnight fast of at least 10 hours, a single oral dose of 140 mg tablet was administered to each participant in a sitting posture with about 240 mL of drinking water in the presence of the principal investigator and quality assurance personnel, and in accordance with the randomization schedule.
  Interventions: Drug: Dasatinib 140 MG [Sprycel]

INTERVENTIONS:
Drug: Dasatinib ASD 100 mg — XS004 Dasatinib Amorphous Solid Dispersion Film-Coated Tablet, 100 mg Test Formulation
  Arms: XS004 - Period 1; XS004 - Period 2; XS004 - Period 3; XS004 - Period 4
Drug: Dasatinib 140 MG [Sprycel] — SPRYCEL® (dasatinib) 140 mg Film-Coated Tablets
  Arms: SPRYCEL - Period 1; SPRYCEL - Period 2; SPRYCEL - Period 3; SPRYCEL - Period 4

SUMMARY:
An open label, single-center, balanced, randomized, two-treatment, two-sequence, four-period, full replicate, crossover, single dose, Phase I, oral comparative bioavailability study in healthy, adult participants (male subjects and female subjects of non-childbearing potential) under fasting conditions with a screening period of 21 days prior to enrollment. In each study period, 21 blood samples were collected from each participant to analyze the pharmacokinetic profile of the test as well as the reference drug.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males (sterile or using contraception) or females of non-childbearing potential 18 and 55 years of age
* Acceptable medical history, physical examination, laboratory investigations within 21 days prior to enrollment
* Clinical laboratory values were within the laboratory's stated normal range. If not within this range, they must be without clinical significance, as determined by the Investigator
* The subject is able to communicate meaningfully with study personnel and is anticipated to be able to comply fully with study procedures

Exclusion Criteria:

* Any history of impairment of cardiovascular, pulmonary, hepatic, renal, gastrointestinal, endocrine, immunological, dermatological, neurological, psychiatric disease or disorder
* Participated in any other clinical study or donated blood in last 90 days
* Positive screens for serum hepatitis B surface antigen (HbsAg), hepatitis C antibody (HepC) or human immunodeficiency virus (HIV)
* Female subjects demonstrating a positive pregnancy screen, currently breastfeeding or using hormone replacement therapy within three months prior to dosing of test product

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 110 (Actual)
Dates: Start 2021-06-07 (Actual); Primary Completion 2021-06-25 (Actual); Study Completion 2021-06-25 (Actual)

PRIMARY OUTCOMES:
Maximum Observed Plasma Concentration (Cmax) of XS004 and SPRYCEL® | For each study period, blood samples were drawn at pre-dose (0.00) and at 0.25, 0.33, 0.50, 0.75, 1.00, 1.25, 1.50, 1.75, 2.00, 2.50, 3.00, 4.00, 5.00, 6.00, 8.00, 12.00, 16.00, 20.00, 24.00, and 30.00 hours post-dose.
  The pharmacokinetic parameters (Cmax) were determined for the test and reference products (XS004 and SPRYCEL®, respectively) for each subject using non-compartmental methods.
Area Under the Plasma Concentration-Time Curve from Zero to the Last Measurable Concentration (AUC0-t) of XS004 and SPRYCEL® | For each study period, blood samples were drawn at pre-dose (0.00) and at 0.25, 0.33, 0.50, 0.75, 1.00, 1.25, 1.50, 1.75, 2.00, 2.50, 3.00, 4.00, 5.00, 6.00, 8.00, 12.00, 16.00, 20.00, 24.00, and 30.00 hours post-dose.
  The pharmacokinetic parameters (AUC 0-t) were determined for the test and reference products (XS004 and SPRYCEL®, respectively) for each subject using non-compartmental methods.
Area Under the Plasma Concentration-Time Curve from Zero Extrapolated to Infinity (AUC0-inf) of XS004 and SPRYCEL® | For each study period, blood samples were drawn at pre-dose (0.00) and at 0.25, 0.33, 0.50, 0.75, 1.00, 1.25, 1.50, 1.75, 2.00, 2.50, 3.00, 4.00, 5.00, 6.00, 8.00, 12.00, 16.00, 20.00, 24.00, and 30.00 hours post-dose.
  The pharmacokinetic parameters (AUC 0-inf) were determined for the test and reference products (XS004 and SPRYCEL®, respectively) for each subject using non-compartmental methods.

SECONDARY OUTCOMES:
Area Under the Plasma Concentration-Time Curve (Percent Extrapolation) of XS004 and SPRYCEL® | For each study period, blood samples were drawn at pre-dose (0.00) and at 0.25, 0.33, 0.50, 0.75, 1.00, 1.25, 1.50, 1.75, 2.00, 2.50, 3.00, 4.00, 5.00, 6.00, 8.00, 12.00, 16.00, 20.00, 24.00, and 30.00 hours post-dose.
  The pharmacokinetic parameters (AUC %Extrap) were determined for the test and reference products (XS004 and SPRYCEL®, respectively) for each subject using non-compartmental methods.
Time of Maximum Observed Plasma Concentration (Tmax) of XS004 and SPRYCEL® | For each study period, blood samples were drawn at pre-dose (0.00) and at 0.25, 0.33, 0.50, 0.75, 1.00, 1.25, 1.50, 1.75, 2.00, 2.50, 3.00, 4.00, 5.00, 6.00, 8.00, 12.00, 16.00, 20.00, 24.00, and 30.00 hours post-dose.
  The pharmacokinetic parameters (Tmax) were determined for the test and reference products (XS004 and SPRYCEL®, respectively) for each subject using non-compartmental methods.
Terminal Half-Life (T1/2) of XS004 and SPRYCEL® | For each study period, blood samples were drawn at pre-dose (0.00) and at 0.25, 0.33, 0.50, 0.75, 1.00, 1.25, 1.50, 1.75, 2.00, 2.50, 3.00, 4.00, 5.00, 6.00, 8.00, 12.00, 16.00, 20.00, 24.00, and 30.00 hours post-dose.
  The pharmacokinetic parameters (T1/2) were determined for the test and reference products (XS004 and SPRYCEL®, respectively) for each subject using non-compartmental methods.
Elimination Rate Constant (Kel) of XS004 and SPRYCEL® | For each study period, blood samples were drawn at pre-dose (0.00) and at 0.25, 0.33, 0.50, 0.75, 1.00, 1.25, 1.50, 1.75, 2.00, 2.50, 3.00, 4.00, 5.00, 6.00, 8.00, 12.00, 16.00, 20.00, 24.00, and 30.00 hours post-dose.
  The pharmacokinetic parameters (Kel) were determined for the test and reference products (XS004 and SPRYCEL®, respectively) for each subject using non-compartmental methods. Apparent first-order terminal elimination rate constant calculated from a semi-log plot of the plasma concentration versus time curve.
Lower Limit on Time for Elimination Rate Constant (Kel_lower) of XS004 and SPRYCEL® | For each study period, blood samples were drawn at pre-dose (0.00) and at 0.25, 0.33, 0.50, 0.75, 1.00, 1.25, 1.50, 1.75, 2.00, 2.50, 3.00, 4.00, 5.00, 6.00, 8.00, 12.00, 16.00, 20.00, 24.00, and 30.00 hours post-dose.
  The pharmacokinetic parameters (Kel_lower) were determined for the test and reference products (XS004 and SPRYCEL®, respectively) for each subject using non-compartmental methods. Apparent first-order terminal elimination rate constant calculated from a semi-log plot of the plasma concentration versus time curve. Kel_lower is the lower limit on time for the elimination rate constant.
Upper Limit on Time for Elimination Rate Constant (Kel_upper) of XS004 and SPRYCEL® | For each study period, blood samples were drawn at pre-dose (0.00) and at 0.25, 0.33, 0.50, 0.75, 1.00, 1.25, 1.50, 1.75, 2.00, 2.50, 3.00, 4.00, 5.00, 6.00, 8.00, 12.00, 16.00, 20.00, 24.00, and 30.00 hours post-dose.
  The pharmacokinetic parameters (Kel_upper) were determined for the test and reference products (XS004 and SPRYCEL®, respectively) for each subject using non-compartmental methods. Apparent first-order terminal elimination rate constant calculated from a semi-log plot of the plasma concentration versus time curve. Kel_upper is the upper limit on time for the elimination rate constant.

CONTACTS AND LOCATIONS:
Overall Officials: Per Andersson, PhD, Study Director — Xspray Pharma AB
Locations (1):
- QPS Bioserve India Pvt Limited, Hyderabad, India

IPD SHARING:
Plan to Share IPD: No